CLINICAL TRIAL: NCT01562964
Title: The Impact of Hypnotherapy on Symptoms, Psychological Morbidity and Quality of Life in Postmenopausal Women With Chest Pain and Unobstructed Coronary Arteries
Brief Title: Hypnotherapy in Patients With Chest Pain & Unobstructed Coronaries
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P40285
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2015-08

CONDITIONS: Chest Pain; Unobstructed Coronary Arteries
MeSH Terms: conditions — Chest Pain | interventions — Hypnosis; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypnotherapy (Experimental): Hypnotherapy will be conducted at the Royal Brompton Hospital by a qualified practician (DF). Ten pain control hypnotherapy session will run for 50-60 minutes each. In the first session a thorough history will be taken of the patient's chest pain history together with both the sensory and affective components of their pain. If there is time, relaxation technique and self-hypnosis will be taught at this visit. In subsequent sessions, various techniques, including techniques that focus on direct suggestions and imagery work, will be applied and taught to the patient. The pain control techniques are all analgesic in nature - focusing on the reduction, but not the total removal of the pain. A small amount of pain is left behind to serve as a reminder that either something is wrong or that the patient needs to take it easy.
  Interventions: Behavioral: Hypnotherapy
- Supportive therapy (Active Comparator): Subjects in the Supportive therapy group will attend the Royal Brompton Hospital weekly for 10 weeks to meet with person of equal status to the hypnotherapist (e.g. a research assistant, not a medical practitioner) trained to provide counseling and support. Visits will last 50-60 min. Patients will be encouraged to talk about their physical symptoms and any emotional issues, and to discuss how these might be coped with in a better way.
  Interventions: Behavioral: Supportive therapy

INTERVENTIONS:
Behavioral: Hypnotherapy — Ten pain control hypnotherapy session will run for 50-60 minutes each. In the first session a thorough history will be taken of the patient's chest pain history together with both the sensory and affective components of their pain. If there is time, relaxation technique and self-hypnosis will be taught at this visit. In subsequent sessions, various techniques, including techniques that focus on direct suggestions and imagery work, will be applied and taught to the patient. The pain control techniques are all analgesic in nature - focusing on the reduction, but not the total removal of the pain. A small amount of pain is left behind to serve as a reminder that either something is wrong or that the patient needs to take it easy.
  Arms: Hypnotherapy
Behavioral: Supportive therapy — Subjects in the Supportive therapy group will attend the Royal Brompton Hospital weekly for 10 weeks to meet with person of equal status to the hypnotherapist (e.g. a research assistant, not a medical practitioner) trained to provide counseling and support. Visits will last 50-60 min.
  Arms: Supportive therapy

SUMMARY:
This study will investigate whether clinical hypnotherapy can effectively treat chest pain symptoms, improve emotional wellbeing and quality of life in postmenopausal women with chest pain and coronary arteries without any narrowings. The diagnosis of chest pain with 'normal' coronary arteries is found in 25% of patients undergoing investigation of chest pain using coronary angiography (when dye is injected into the coronary arteries whilst xray pictures are taken), and the majority of these patients are postmenopausal women. Often there is no obvious physical cause. Despite symptoms being treated using conventional drugs, and life expectancy is not affected, many patients continue to suffer from debilitating chest pain symptoms, frequently resulting in visits to hospital, increased psychological illness and poor quality of life. The investigators are interested in finding ways of improving not only chest pain symptoms but also psychological wellbeing and quality of life in these patients. Previous studies of ours have found improvement in these patients after taking part in a support group, and using a relaxation technique called Autogenic training. Recently the investigators conducted a pilot study which showed a favourable effect of hypnotherapy on physical ability, well-being and quality of life. The investigators would now like to extend this study, performing a larger randomised, controlled trial. The investigators hypothesise that hypnotherapy will beneficially affect symptoms and quality of life in patients with cardiac Syndrome X.

ELIGIBILITY:
Inclusion Criteria:

* history of chest pain for ≥ 2 years
* ≥ 2 episodes chest pain per week
* angiographically smooth epicardial coronary arteries
* Willing to give written informed consent

Exclusion Criteria:

* Any epicardial coronary atheroma on angiography of the coronary arteries
* left ventricular hypertrophy or dysfunction (clinical/ECG/echo/CXR)
* previous hypnotherapy for chest pain symptoms
* participation in research project within previous 60 days
* unwilling to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2012-03-02 (Actual); Study Completion 2012-03-02 (Actual)

PRIMARY OUTCOMES:
Symptom frequency | 24 weeks

SECONDARY OUTCOMES:
Symptom severity | 24 weeks
Psychological morbidity | 24 weeks
General quality of life | 24 weeks
  Using Short Form 36 questionnaire
Hospitalisations | 24 weeks
Consultancy time | 24 weeks
Medication use | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Collins, MD, FRCP, Principal Investigator — Imperial College London, and Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton & Harefield NHS Foundation Trust, London, United Kingdom